CLINICAL TRIAL: NCT00449085
Title: Clinical Evaluation of the CARTO™ XP EP Navigation System v9 and Biosense Webster SOUNDSTAR 3D Diagnostic Ultrasound. A Feasibility Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Collaborators: Royal Adelaide Hospital (Other); Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RAH061225
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Electrophysiology
Device: CARTO™ XP EP Navigation System V9

SUMMARY:
Feasibility study to evaluate CARTO™ XP EP Navigation System V9 and SOUNDSTAR 3D Diagnostic Ultrasound Catheter.

DETAILED DESCRIPTION:
To construct geometric representation of the heart chambers using intracardiac ultrasound.The Carto™ XP Electrophysiology (EP) Navigation System v9 is intended to acquire real-time catheter based cardiac electrophysiogical maps.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing any EPS study and or Ablation will be eligible for this study.

Age 18 years or older Signed Patient Informed Consent Form

Exclusion Criteria:

* Patients with inadequate vascular access

Patients with any of the following criteria will be excluded:

* Women who are pregnant

  * Age <18 years
  * Any Contraindication to the clinical procedure
  * Sepsis
* Major coagulation abnormalities
* Presence of any intracardiac thrombus
* Unstable angina
* Uncontrolled Heart failure
* Deep Vein Thrombosis
* Significant peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prashanthan Sanders, MBBS,PhD,FRCACP, Study Director — Royal Adelaide Hospital; Jonathan Kalman, MBBS,PhD,FRACP, Principal Investigator — Melbourne Health